CLINICAL TRIAL: NCT00005455
Title: Chagas Disease as an Undiagnosed Type of Cardiomyopathy in the United States
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4488; Z01HL005264 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2001-11

CONDITIONS: Heart Diseases; Myocardial Diseases; Chagas Disease
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies; Chagas Disease

SUMMARY:
A detailed review was made of data pertinent to the occurrence of chronic Chagas disease in the United States.

DETAILED DESCRIPTION:
BACKGROUND:

In Latin America, 16 to 18 million individuals are thought to have Chagas' disease and 90 million are considered to be at risk of infection. In the United States, the occurrence of Chagas' disease is virtually limited to individuals who have resided in Latin America where they acquired the infection, and then migrated to this country.

DESIGN NARRATIVE:

Data on the prevalence of positive serologic reactions for Trypanosoma cruzi (a protozoan causing Chagas cardiomyopathy) serve for calculating that a total of up to 74,000 Latin Americans residing in the United States have the chronic form of chagasic cardiomyopathy. The vast majority of these individuals are either undiagnosed, or misdiagnosed as having idiopathic dilated cardiomyopathy or coronary artery disease. Vector transmission of T. cruzi infection is very unlikely to occur in the United States because of variations in biological behavior of local species of insect vectors and because of changes in human living conditions. Transfusion of blood from infected but asymptomatic individuals is considered the most important mechanism of transmission of this disorder in the United States.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-01; Study Completion 1993-12 (Actual)